CLINICAL TRIAL: NCT06497543
Title: The Efficacy and Safety of Intrathecal Pemetrexed for SCLC Patients With Refractory Brain Metastases or Leptomeningeal Metastasis: A Phase II Study
Brief Title: Intrathecal Pemetrexed for SCLC Patients With Refractory Brain Metastases or Leptomeninges Metastatic
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Collaborators: Second People's Hospital of Hunan (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Head of Medical Oncology, Director of Early Clinical Trial Center, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240705
Record Dates: First submitted 2024-07-05; First posted 2024-07-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Small Cell Lung Cancer patient with Refractory Brain Metastases
  Interventions: Drug: Intrathecal Pemetrexed
- Cohort 2 (Experimental): Small Cell Lung Cancer patient with Leptomeningeal Metastasis
  Interventions: Drug: Intrathecal Pemetrexed

INTERVENTIONS:
Drug: Intrathecal Pemetrexed — Intrathecal pemetrexed(50mg) twice a week for 1 week (day 1 and day 5) as induction treatment, then once monthly until progressive disease.
  Other Names: Pemetrexed

SUMMARY:
This study aimed to evaluate the efficacy and safety of intrathecal pemetrexed for SCLC patients with refractory brain metastases or leptomeningeal metastasis.

DETAILED DESCRIPTION:
This is a prospective interventional clinical study to evaluate the efficacy and safety of intrathecal pemetrexed for SCLC patients with refractory brain metastases or leptomeningeal metastasis. Approximately 80 small cell lung cancer patients with refractory brain and/or leptomeningeal metastasis were enrolled and treated with intrathecal pemetrexed, there were 40 cases in cohort 1 with refractory brain metastasis and 40 cases in cohort 2 with leptomeningeal metastasis.Cerebrospinal fluid samples will be collected before and after pemetrexed resistance to analyze molecular mechanisms. The study is expected to commence recruitment in mainland China in about September 2024. It is expected that the trial will end in April 2026.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understand the requirements and contents of the clinical trial, and provide a signed and dated informed consent form.
* 2. Age ≥ 18 years.
* 3. Histopathology is confirmed small cell lung cancer .
* 4.Leptomeningeal metastasis (LM) is defined by the presence of typical clinical symptoms, positive cerebrospinal fluid (CSF) cytology, detection of cell-free DNA (cfDNA) in CSF by next-generation sequencing (NGS), or imaging findings consistent with typical meningeal metastases.
* 5.Patients with brain progression after whole-brain radiotherapy.
* 6. Predicted survival ≥ 12 weeks. .
* 7. ECOG 0-2.
* 8. Adequate bone marrow hematopoiesis and organ function.

Exclusion Criteria:

* 1. Previously received intrathecal pemetrexed therapy for locally advanced or metastatic disease.
* 2. Subjects who have received any of the following treatments must be excluded:
* Have received radiation within 14 days prior to the first dose or have not recovered from radiation-related toxicity. Chest and extra-brain palliative radiotherapy, stereotactic radiosurgery, and stereotactic body radiotherapy may be performed 7 days prior to the first dose.
* 3. Presence of spinal cord compression or meningeal metastasis.
* 4. History of other malignant tumors within 2 years.
* 5. Adverse events (except alopecia of any degree) of CTCAE > grade 1 due to prior treatment (e.g., adjuvant chemotherapy, radiotherapy, etc.) prior to the first dose.
* 6. History of stroke or intracranial hemorrhage within 6 months prior to the first dose.
* 7. The presence of any severe or poorly controlled systemic disease, including poorly controlled hypertension and active bleeding in the judgment of the investigator.
* 8. Subjects with persistent or active infection, including but not limited to hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) and COVID-19 infection.
* 9. Heart-related diseases or abnormalities
* 10. Past history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy or interstitial lung disease with active clinical symptoms, immune pneumonia caused by immunotherapy.
* 11. Refractory nausea and vomiting, chronic gastrointestinal disease, difficulty swallowing drugs, or inability to adequately absorb sunvozertinib or anlotinib due to previous bowel resection.
* 12. Live vaccine was given 2 weeks before the first medication.
* 13. Women who are breastfeeding or pregnant.
* 14. Hypersensitivity to the test drug and the ingredients.
* 15. Other conditions assessed by the investigator to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Time from first subject dose to study completion, or up to last follow up
  OS was defined as the duration from the start of intrathecal pemetrexed to patient death

SECONDARY OUTCOMES:
Intracranial progression-free survival (I-PFS) | Time from first subject dose to study completion, or up to 36 month
  Intracranial progression-free survival was defined as the duration from the start of intrathecal pemetrexed to the worsening of neurological symptoms, radiological confirmation of brain progression, or patient death
Intracranial Objective Response Rate (I-ORR) | Time from first subject dose to study completion, or up to 36 month
  To assess Intracranial overall response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as the proportion of subjects who have a complete response (CR) or a partial response (PR)
clinical remission rate | Time from first subject dose to study completion, or up to 36 month
  Clinical Response Rate was defined as the ratio of the patient whose neurological symptoms and KPS improved according to the criteria of clinical response
Adverse events (AEs) | Time from first subject dose to study completion, or up to 36 month
  Number of participants with adverse events (AEs) according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Yongchang Zhang, Changsha, Hunan, China